CLINICAL TRIAL: NCT07082452
Title: A Randomized, Open-labelled, Multicenter Trial Evaluating Efficacy and Safety of A Reduced Venetoclax Exposure To Seven Days Versus Standard Continuous Venetoclax Exposure Combined With Azacitidine in Treatment Naïve Subjects With Acute Myeloid Leukemia Who Are Ineligible for Intensive Induction
Brief Title: A Multicenter Trial Evaluating Efficacy and Safety of A Reduced Venetoclax Exposure To Seven Days Versus Standard Continuous Venetoclax Exposure Combined With Azacitidine in Treatment Naïve Subjects With Acute Myeloid Leukemia Who Are Ineligible for Intensive Induction
Acronym: SEVENAZA
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-521634-29-00; 2025-521634-29-00 (EU CTIS Number); 2025/4132 (Other: CSET number (Gustave Roussy ID))
Record Dates: First submitted 2025-06-23; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Leukemia, B-Cell, Chronic; Leukemia
Keywords: Acute Myeloid Leukemia, Venetoclax Exposure, Venetoclax, Azacitidine
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia; Leukemia, Myeloid, Acute | interventions — venetoclax; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Venetoclax (7 days) + Azacitidine (Experimental): Arm A (experimental): Patients will receive venetoclax for a total of seven days.
  * Azacitidine 75 m Subcutaneous (SC) or intravenous (IV) Daily with a continuous 7-day scheme or on a 5-on/2-off [weekend]/2-on schedule (5-0-2) in 28-day cycle
  * Venetoclax 400 mg orally once Daily on Days 1 - 7, in case of AZA treatment with a continuous 7-day scheme OR Venetoclax 400 milligram (mg) Daily on Days 1 - 5 and Day 8-9 in case of AZA treatment with a 5-0-2 scheme.
  Interventions: Drug: Venetoclax; Drug: Azacitidine
- Arm B: Venetoclax (28 days) + Azacitidine (Active Comparator): Arm B (standard): Patients will receive venetoclax for a total of 28 days (before remission), according to VIALE-A protocol.
  * Azacitidine 75 mg/m2 Subcutaneous (SC) or IV Daily with a continuous 7-day scheme or on a 5-on/2-off [weekend]/2-on schedule (5-0-2) in 28-day cycle.
  * Venetoclax 400 mg orally once Daily on Days 1 - 28.
  Interventions: Drug: Venetoclax; Drug: Azacitidine

INTERVENTIONS:
Drug: Venetoclax — Venetoclax 400 mg orally once Daily
Drug: Azacitidine — 75 mg/m2 Subcutaneous (SC) or intravenous (IV) Daily with a continuous 7-day scheme or on a 5-on/2-off [weekend]/2-on schedule (5-0-2) in 28-day cycle

SUMMARY:
Combination of azacitidine (AZA) for 7 days every 28 days with a continuous daily exposure to Venetoclax (VEN), an oral bcl-2 inhibitor, is now approved for the treatment of acute myeloid leukemia (AML) in patients ineligible for intensive chemotherapy due to age (>75 years) or comorbidities. VEN+AZA showed significant overall response rate and survival benefit but combination carries a risk of considerable toxicity (such as profound/prolonged cytopenia and infections) before but also after remission. These toxicities make it difficult to apply the recommended treatment regimen, in particular the continuous daily intake of VEN. Recent reports suggest that reducing VEN duration per cycle seems safe and feasible. We propose to investigate a reduced-intensity VEN regimen (7-day dosing/28) versus the standard continuous VEN therapy (28-day dosing/28), combined with AZA, with the primary goal of maintaining efficacy while reducing associated toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have confirmation of AML by WHO 2022 criteria and be ineligible for treatment with a standard cytarabine and anthracycline induction regimen due to age or co-morbidities.
2. Subject must be ≥ 60 years of age.
3. Subject must have a projected life expectancy of at least 12 weeks.
4. Subject must be considered ineligible for induction therapy defined by the following:

   * 75 years of age OR
   * 60 to 74 years of age with at least one of the following co-morbidities:

     * ECOG Performance Status of 2 or 3;
     * Cardiac history of CHF requiring treatment or Ejection Fraction ≤ 50% or chronic stable angina;
     * DLCO ≤ 65% or FEV1 ≤ 65%;
     * Severe Renal impairment: Creatinine clearance ≥ 30 mL/min to < 45 ml/min
     * Moderate hepatic impairment with total bilirubin > 1.5 to ≤ 3.0 × ULN
     * Any other comorbidity that the physician judges to be incompatible with intensive chemotherapy must be reviewed and approved by the coordinator before study enrollment
5. Subject must have an Eastern Cooperative Oncology Group (ECOG) Performance status (Appendix 4):

   * 0 to 2 for subject ≥ 75 years of age.
   * 0 to 3 for subject ≥ 60 to 74 years of age.
6. Subject must have adequate renal function as demonstrated by a creatinine clearance ≥ 30 mL/min; calculated by the Cockcroft Gault formula.
7. Subject must have adequate liver function as demonstrated by:

   * Aspartate aminotransferase (AST) ≤ 3.0 × ULN*
   * Alanine aminotransferase (ALT) ≤ 3.0 × ULN*
   * Bilirubin ≤ 1.5 × ULN*.

   (* Unless considered to be due to leukemic organ involvement. Subjects who are < 75 years of age may have a bilirubin of ≤ 3.0 × ULN)
8. Female subjects must be either postmenopausal (amenorrhea for at least 12 months with no alternative medical reasons) or surgically sterile (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
9. Non-sterile male subjects must use contraceptive methods with partner(s) prior to beginning study drug administration and continuing up to 90 days after the last dose of study drug. Male subjects must agree to refrain from sperm donation from initial study drug administration until 90 days after the last dose of study drug.
10. Subject must voluntarily sign and date an informed consent, approved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB), prior to the initiation of any screening or study specific procedures.
11. Patients must be affiliated to a social security system or beneficiary of the same
12. Patients shall be eligible to undergo Azacitidine and Venetoclax treatment and BM aspiration. Patients who either do not consent to a BM aspiration will not be eligible.

Exclusion Criteria:

1. Subject has received treatment with the following:

   * Hypomethylating agent, venetoclax and/or any chemo-therapeutic agent for Myelodysplastic syndrome (MDS).
   * Chimeric Antigen Receptor (CAR)-T cell therapy.
   * Experimental therapies for MDS or Acute Myeloid Leukemia (AML).
   * Current participation in another research or observational study.
2. Subject has history of myeloproliferative neoplasm [MPN], including myelofibrosis, essential thrombocythemia, polycythemia vera, chronic myeloid leukemia (CML) with or without BCR-ABL1 translocation and AML with BCR-ABL1 translocation.
3. Subject has favorable risk cytogenetics such as t(8;21), inv(16), t(16;16) or t(15;17) as per the NCCN Guidelines Version 2, 2016 for Acute Myeloid Leukemia.
4. Subject has acute promyelocytic leukemia
5. Subject has known active CNS involvement with AML.
6. Known human immunodeficiency virus HIV
7. Known hepatitis B or C infection with the exception of those with an undetectable viral load within 3 months.
8. Subject has a cardiovascular disability status of New York Heart Association Class ≥ 2. Class 2 is defined as cardiac disease in which patients are comfortable at rest but ordinary physical activity results in fatigue, palpitations, dyspnea, or anginal pain.
9. Subject has chronic respiratory disease that requires continuous oxygen, or significant history of renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic, hepatic, cardiovascular disease, or any other medical condition that in the opinion of the investigator would adversely affect his/her participating in this study.
10. Subject has a malabsorption syndrome or other condition that precludes enteral route of administration.
11. Subject exhibits evidence of other clinically significant uncontrolled systemic infection requiring therapy (viral, bacterial or fungal).
12. Subject has a history of other malignancies prior to study entry, with the exception of:

    * Adequately treated in situ carcinoma of the cervix uteri or carcinoma in situ of breast;
    * Basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin;
    * Previous malignancy confined and surgically resected (or treated with other modalities) with curative intent and considered in remission for 3 years.
13. Subject has a white blood cell count > 25 × 109/L. (Hydroxyurea is permitted to meet this criterion.)
14. Subject has hypersensitivity to the active substances of any of the excipients
15. Patient under guardianship or deprived of his liberty by a judicial or administrative decision or incapable of giving its consent

NB: patients with IDH1-mutant AML will not be formally excluded from the study. However, investigators are strongly encouraged to prefer treatment combining Azacitidine and Ivosidenib (AGILE phase III trial).

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 262 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2030-09 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with complete remission or complete remission with incomplete marrow recovery (CR/CRi) | at any time point during the study (at 30 days, 60 days, 3 years)
  This proportion will be calculated based on current IWG criteria for AML

SECONDARY OUTCOMES:
Overall survival (OS) | at 30 days, 60 days, 1, 2 and 3 years
Event-Free Survival (EFS) | at 30 days, 60 days, 1, 2 and 3 years
  Defined as the number of days from the date of randomization to the date of treatment failure, hematologic relapse from CR/CRh/CRi or death from any cause, whichever occurs first.
Early mortality rate | At day 60
Time to first response | at 30 days, 60 days, 1, 2 and 3 years
  Defined as the number of days from the date of randomization to the date of earliest CR or CRi
Time to best response | at 30 days, 60 days, 1, 2 and 3 years
  Defined as the number of days from the date of randomization to the date of CR (or CRi if patients never reached CR).
Duration of response (DoR) | at 30 days, 60 days, 1, 2 and 3 years
  Among subjects who achieved CR and CRi, duration of response (DOR) will be calculated as the date of the first response to the date of first documented disease relapse, disease progression, treatment failure, or death.
Venetoclax (VEN) scheme modification (dosing schedule modification, delays >2 days or discontinuation) | until the last cycle of treatment (up to 3 years)
  Defined as the proportion of CR/CRi patients that presented treatment modification not authorized by protocol as VEN schedule modification (dose, duration), delay >2 days from the initial Day of the subsequent cycle and/or temporary/definitive VEN discontinuation.
Platelet transfusion requirement | At 24 weeks
  measured by the number of platelet concentrates received by patient during each cycle from cycle 1 day 1 to relapse or last day of cycle 6.
Febrile neutropenia or severe infection (grade III/IV) incidence | At 24 weeks
  measured by the number of episodes of febrile neutropenia or severe infection (grade III/IV) by patient during each cycle from cycle 1 day 1 to relapse or last day of cycle 6.
Hospitalization requirement and length stay | At 24 weeks
  Hospitalization requirement will be defined as number of all hospitalization longer than 24h during each cycle from Cycle 1 Day 1 to relapse or last day of Cycle 6. Hospitalization length stay will be defined by the addition of number of days of each hospitalization longer than 24h during each cycle from cycle 1 day 1 to relapse or last day of cycle 6.

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy, Villejuif, France

IPD SHARING:
Plan to Share IPD: No